CLINICAL TRIAL: NCT06544460
Title: Secondary Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy for Recurrent Ovarian Cancer Patients With PARP Inhibitors Resistance: a Phase II Clinical Study
Brief Title: Secondary Cytoreduction and Hyperthermic Intraperitoneal Chemotherapy for PARP Inhibitors Resistance Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Director of Gynecological Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OCR-HIPEC-2024
Record Dates: First submitted 2024-07-29; First posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; hyperthermic intraperitoneal chemotherapy; secondary cytoreduction
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Recurrent Ovarian Cancer After PARPi Therapy (Experimental): After treated with PARP inhibitors, patients have recurrent ovarian cancer and need a surgery.
  Interventions: Procedure: Secondary cytoreduction; Drug: Hyperthermic intraperitoneal chemotherapy

INTERVENTIONS:
Procedure: Secondary cytoreduction — Repeated tumor cell reduction surgery for recurrent ovarian cancer patients
Drug: Hyperthermic intraperitoneal chemotherapy — Using the BR-TQR-I intraperitoneal hyperthermic perfusion chemotherapy instrument, after the surgical operation is completed, four drainage tubes are placed in the left and right upper abdomen and lower abdomen respectively. Connect all pipelines and preheat the instrument before starting treatment. The treatment temperature is controlled at 43 ℃± 0.1 ℃, the treatment time is 90 minutes, and the circulation pump flow rate is 400-600ml/min. Within 48 hours after the surgery, cisplatin 75mg/㎡ was added to 3000ml of physiological saline for intraperitoneal hot infusion. Through the comprehensive effects of circulation flushing, hyperthermia, chemotherapy, and thermochemotherapy sensitization, it kills and removes residual cancer cells or small lesions in the abdominal cavity.

SUMMARY:
At present, the treatment of recurrent ovarian cancer after PARP inhibitor therapy is quite challenging, and there is no research on the application of hyperthermic intraperitoneal chemotherapy(HIPEC) for the above-mentioned patients. Therefore, this study aims to explore the safety and efficacy of secondary cytoreduction combined with hyperthermic intraperitoneal chemotherapy for recurrent ovarian cancer after maintenance therapy with PARP inhibitors through a single-center, prospective, single-arm, phase II clinical trial. The goal is to explore the treatment options for ovarian cancer patients in the era of PARP inhibitors, thereby improving the overall treatment level and prognosis of ovarian cancer.

DETAILED DESCRIPTION:
1. Overall design This is a single-center, prospective, single-arm, phase II clinical trial to evaluate the safety and efficacy of decellularization combined with intraperitoneal hyperthermic perfusion for recurrent ovarian cancer after maintenance therapy with PARP inhibitors.
2. Sample size calculation This clinical trial aims to evaluate the safety and efficacy of decellularization combined with intraperitoneal hyperthermic perfusion for the maintenance treatment of recurrent ovarian cancer with PARP inhibitors. The median progression-free survival of patients who received maintenance therapy with PARP inhibitors in our center is 11 months. It is expected that HIPEC can reduce the risk of recurrence by 30%. After 1 year of enrollment and 2 years of follow-up, the alpha value is 0.05. Considering the participants who withdrew from the study midway or dropped out due to loss to follow-up, this study intends to include 94 participants.
3. Methods Using the BR-TQR-I intraperitoneal hyperthermic perfusion chemotherapy instrument, after the surgical operation is completed, four drainage tubes are placed in the left and right upper abdomen and lower abdomen respectively. Connect all pipelines and preheat the instrument before starting treatment. The treatment temperature is controlled at 43 ℃± 0.1 ℃, the treatment time is 90 minutes, and the circulation pump flow rate is 400-600ml/min. Within 48 hours after the surgery, cisplatin 75mg/㎡ was added to 3000ml of physiological saline for intraperitoneal hot infusion.
4. Data statistics Enter data and use SPSS statistical software for statistical analysis. Statistical analyst: Clinical Statistics Department of Fudan University Cancer Hospital. Mailing address: 270 Dong'an Road, Shanghai.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with previously diagnosed ovarian cancer, fallopian tube cancer, or primary peritoneal cancer;
2. Maintain treatment with PARP inhibitors before recurrence;
3. The imaging assessment is suitable, and the patient agrees to undergo further cytoreductive surgery;
4. The outcome of recurrent surgery is R0 or R1 resection;
5. Sign the informed consent form;
6. Age≥18 years old;

Exclusion Criteria:

1. Patients with ovarian cancer excluded by pathological or clinical diagnosis;
2. Inappropriate imaging evaluation or physical intolerance for surgical patients;
3. Isolated lymph node recurrence
4. Patients who undergo unsatisfactory tumor reduction surgery (R2 resection) due to recurrence;
5. Patients who are unwilling to participate in the clinical trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2024-08-31 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
PFS | Two years
  Progression free survival

SECONDARY OUTCOMES:
OS | Two years
  Overall Survival

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan university shanghai cancer center, Deparment of gynecologic oncology, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No